CLINICAL TRIAL: NCT04853784
Title: Prospective Registration Study of Totally Laparoscopy Versus Laparoscopy Assisted Colon Cancer Surgery
Acronym: STARS-CC01
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Professor, The First Hospital of Jilin University
Other Study IDs: STARS-CC01
Record Dates: First submitted 2021-04-06; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Colon Cancer; Surgery; Totally Laparoscopic; Intracorporeal Anastomosis
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Totally laparoscopic colon surgery: Totally laparoscopic colon surgery/intracorporeal anastomosis
  Interventions: Procedure: intracorporeal anastomosis
- Laparoscopic-assited colon surgery: Laparoscopic-assited colon surgery/extracorporeal anastomosis
  Interventions: Procedure: intracorporeal anastomosis

INTERVENTIONS:
Procedure: intracorporeal anastomosis — intracorporeal anastomosis
  Other Names: extracorporeal anastomosis

SUMMARY:
This is a comparison of totally laparoscopic and laparoscopic-assisted colon cancer resection, a prospective registration study comparing the safety and benefits of the two operations

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common malignant tumors in China. With the advancement of medical science and technology, the treatment of colorectal cancer has become more mature, forming a comprehensive and individualized treatment model focusing on surgery. The promotion of the principles of TME and CME surgery has greatly standardized the operation of colorectal surgery. COLOR II, COREAN and CLASICC studies have all confirmed the safety and effectiveness of laparoscopic colorectal cancer surgery.

In traditional laparoscopic-assisted surgery, a small incision in the abdominal wall is used to assist in trimming the mesangium to remove the specimen, and the anastomosis is completed outside the abdominal wall, which will still cause postoperative incision pain and may lead to complications such as incisional infection and incisional hernia. However, in some obese patients, the mesangium is thick and short. The above operations are more difficult, and may even cause the risk of mesangial tears and bleeding, which will weaken the minimally invasive advantages of laparoscopic surgery.

The total laparoscopic radical resection of colon cancer is performed under laparoscopic free dissection and dissected reconstruction of the operation area. The small incision of the abdominal wall Trocar is used to take out the specimen, which not only guarantees a sufficient range of dissection and resection, but also avoids the troubles caused by the auxiliary abdominal wall incision. Postoperative recovery may be faster, but it also raises questions about the increased risk of infection in the surgical area. Total laparoscopic radical resection of colon cancer still lacks corresponding high-quality clinical research. In response to this problem, this study compares related surgical methods, verifies the safety and effectiveness of the corresponding surgical methods, and provides better guidance for subsequent clinical practice.

Taking laparoscopic-assisted radical resection of colon cancer as a control, the short-term and long-term effects of full laparoscopic radical resection of colon cancer were evaluated, so as to choose a more effective and safe operation method.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old, male or female;
2. Colon cancer (ascending colon, transverse colon, descending colon, sigmoid colon) is diagnosed by histology or cytology;
3. The clinical stage is T1-4aN0-2M0; 4 No multiple distant metastases;

5. ECOG score 0-2; 6. Heart, lung, liver, and kidney functions can tolerate surgery; 7. Patients and their families can understand and are willing to participate in this clinical study, and sign an informed consent.

Exclusion Criteria:

1. Past history of malignant colorectal tumors or recent diagnosis combined with other malignant tumors;
2. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. who need emergency surgery;
3. Neighboring organs need to be combined with organ resection;
4. New adjuvant therapy before surgery;
5. ASA grade ≥ grade IV and/or ECOG physical status score> 2 points;
6. Those who have severe liver and kidney function, cardiopulmonary function, blood coagulation dysfunction, or combined with serious underlying diseases that cannot tolerate surgery;
7. History of severe mental illness;
8. Pregnant or lactating women;
9. Patients with other clinical and laboratory conditions considered by the investigator should not participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complications | 30 days after operation
  Complication incidence 30 days after operation

SECONDARY OUTCOMES:
Operation time | one hour after surgery
  the length between the beginning and the end of the whole operation
number of lymphnodes dissected | During the operation
  one week after surgery
Length of surgical incision | one week after surgery
  Length of surgical incision
Intraoperative blood loss | one hour after surgery
  the mount of blood loss during the whole operation(ml）
Intraoperative conversion rate | one hour after surgery
  Intraoperative conversion rate (conversion to open, conversion to laparoscopic-assisted surgery
Rate of complete mesentery resection (CME) | one week after surgery
  Rate of complete mesentery resection (CME)
Postoperative recovery | During the postoperative hospital stay
  Postoperative recovery: first exhaust, defecation time, restoring liquid diet, hospitalization days.
3-year disease-free survival | 3 years after operation
  3-year disease-free survival
5-year overall survival OS | 5 years after operation
  5-year overall survival OS

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin University First Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No